CLINICAL TRIAL: NCT05490212
Title: Salivary Profiling in Infants Treated for Suspected Sepsis: The SPITSS Study
Acronym: SPITSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tufts Medical Center (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other); University of Florida (Other); Brigham and Women's Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13372
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Infection; Newborn
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples will be obtained every time an infant's caregivers believe the infant is at risk for an infection and the infant is given antibiotics. Saliva will be collected at the beginning of antibiotic treatment; and 2) 18-36 hours into therapy with antibiotics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Single Molecule Array (SiMoA) — The Single Molecule Array (SiMoA), capable of quantifying multiple salivary cytokines from a single sample source at a femtoscale level. The SiMoA platform has been adapted to detect up to nine inflammatory biomarkers, including CRP, PCT, tumor necrosis factor α (TNF α) and ILs 1ß, 6, and 8 in neonatal saliva.

SUMMARY:
The aim of this study is to develop a faster, safer, and more accurate method for determining if a newborn has an infection. This study involves analyzing saliva for markers of infection and inflammation known as cytokines. We will analyze infant's saliva repeatedly for inflammatory biomarkers (cytokines) within the first 36 hours of their standard of care treatment. We hypothesize that levels of these cytokines will more quickly predict which babies are truly infected and which babies are not compared to the blood tests currently being used.

DETAILED DESCRIPTION:
Specific Aim 1: Develop a predictive model of neonatal infection based upon the expression profile of six salivary inflammatory biomarkers, CRP, procalcitonin, tumor necrosis factor-alpha (TNF-α), and interleukins (IL) 1β, 6, and 8, within the first 36 hours of treatment. Serial saliva samples collected at the initiation of antibiotic therapy and 18-36 hours into treatment from 2,250 neonatal 'rule out sepsis' evaluations will undergo multiplexed quantification of the six salivary inflammatory biomarkers. Diagnostic accuracy will be calculated and predictive models will be developed, incorporating clinical, demographic, and biomarker data.

Specific Aim 2: Validate the predictive model of neonatal infection developed in Aim 1 on an external cohort of newborns. Serial saliva samples from an additional, prospective cohort of 1,750 infants undergoing a 'rule out sepsis' evaluation will be collected to test the validity of the predictive model for neonatal infection.

Specific Aim 3: Establish normative salivary reference ranges of the inflammatory biomarkers across varying gestational ages and weights, and assess the potential of these biomarkers to predict other neonatal morbidities. Salivary samples from the subset of uninfected newborns from Aims 1 and 2 will be combined and used to establish the 95% reference intervals of the salivary inflammatory biomarkers at each time point. Salivary profiles will be correlated to discharge diagnoses (i.e. bronchopulmonary dysplasia, periventricular leukomalacia) to assess the ability of each biomarker, alone and in combination, to predict neonatal morbidities known or hypothesized to be associated with an inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

Neonates < 43 weeks' gestation, currently admitted to the NICU or well-baby nursery.

Exclusion Criteria:

Neonates suffering from a lethal genetic or chromosomal abnormality or other non-infectious, life-limiting illness, known at the time parents would be approached for consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Neonates < 43 weeks' gestation, currently admitted to the NICU or well-baby nursery, who undergo a rule-out sepsis evaluation and are started on antibiotics.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-10-03 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
confirmed (culture positive) infection | at initiation-of-rule-out, at 18-to-36-hour, and change between these time points

SECONDARY OUTCOMES:
confirmed (culture positive) infection or clinical infection | at initiation-of-rule-out, at 18-to-36-hour, and change between these time points

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Women and Infants' Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set will be submitted to NIH.